CLINICAL TRIAL: NCT07400380
Title: Prosthetic Complications and Patient Satisfaction of Two Different Implant Distribution for Stress Free Implant Bar Mandibular Overdenture:
Brief Title: Prosthetic Complications and Patient Satisfaction of Two Different Implant Distribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A09011122
Record Dates: First submitted 2026-01-31; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Patient Satisfaction; Prosthetic Complication
Keywords: implant overdenture; bar attachment; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Group 1: four implants were distributed in interforaminal distance, 2-Implant were inserted in canine region and 2-implant 8mm posterior to canine implants.
  Group 2: four implants were distributed in quadrilateral distribution, 2-Implant in canine region and 2-Implant were inserted 26mm posterior to canine implant.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- quadrilateral group (Other): 4-implants were distributed in quadrilateral distribution, 2-Implant in canine region and 2-Implant were inserted 26mm posterior to canine implant.
  Interventions: Procedure: four implants inserted in the mandible and distributed in quadrilateral manner and SFI-Bar had been inserted
- curved group (Other): Receive four implants distributed in interforaminal distance, 2-Implant were inserted in canine region and 2- implant 8mm posterior to canine implants.
  Interventions: Procedure: four implants inserted in the mandible and distributed in quadrilateral manner and SFI-Bar had been inserted

INTERVENTIONS:
Procedure: four implants inserted in the mandible and distributed in quadrilateral manner and SFI-Bar had been inserted — Implant positions were planned at canines for both groups. (Intraforaminal): posterior implants are 8 mm posterior to the canine implants [minimum allowed inter-implant distance for SFIbars (Quadrilateral): posterior implants are 26 mm posterior to the canine implants [Maximum allowed inter-implant distance for SFI-bars
  Other Names: four implants inserted in the mandible and distributed in curved manner and SFI-Bar had been inserted

SUMMARY:
Purpose: This clinical study aimed to evaluate patient satisfaction and prosthetic complications of different distributions of four implants supported mandibular overdentures using Stress free implant bar (SFI-Bar attachments). Evaluation was done for patient satisfaction and prosthetic complications

DETAILED DESCRIPTION:
Purpose: This clinical study aimed to evaluate patient satisfaction and prosthetic complications of different distributions of four implants supported mandibular overdentures using Stress free implant bar (SFI-Bar attachments). Materials and Methods: thirty completely edentulous patients with insufficient retention and stability of their conventional mandibular denture were eligible for this study. All patients received new maxillary and mandibular dentures. The patients were randomly divided into three groups. (G1): four implants were distributed in interforaminal distance, 2-Implant were inserted in canine region and 2- implant 8mm posterior to canine implants. (G2): 4-implants were distributed in quadrilateral distribution, 2-Implant in canine region and 2-Implant were inserted 26mm posterior to canine implant. Patient satisfaction was evaluated by visual analogue scale and prosthetic complications were evaluated on the patient level and implant patients.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of Angel's class I maxillo-mandibular relation.

Exclusion Criteria:

uncontrolled diabetes osteoporosis

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | one year
  A visual analog scale (VAS) and oral health-related quality of life (OHRQoL) were used for evaluating patient satisfaction. Participants in the VAS were instructed to draw a vertical line anywhere along a horizontal line that was used as a scale, with 0 mm representing the worst and 100 mm representing the best. at the point that most accurately reflected their perceptions. General satisfaction, denture stability and retention, occlusion, comfort, ease of cleaning, ease of speaking, ease of chewing, bolus quality, and aesthetics

SECONDARY OUTCOMES:
prosthetic complications | one year
  The complications include (1) complications of attachments: abutment fracture, abutment screw loosening, screw fracture, wear/distortion of retentive components, activation of retentive components, retention loss and replacement of retentive components, and separation of retentive components from the denture base, (2) technical complications of mandibular over-dentures: reline, fracture/remake, teeth wear, teeth separation/fracture, (3) technical complications of maxillary dentures: reline, fracture/remake, teeth wear, teeth separation/fracture, (4) Soft tis-sue complications of mandibular overdentures and maxillary dentures: mucositis, soreness, ulcer decubitus, hyperplasia, and flabbyridge

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Aboelez, profesor, Study Chair — Mansoura University
Locations (1):
- Marwa, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahanna FF, Elsyad MA, Mourad SI, Abozaed HW. Satisfaction and Oral Health-Related Quality of Life of Different Attachments Used for Implant-Retained Overdentures in Subjects with Resorbed Mandibles: A Crossover Trial. Int J Oral Maxillofac Implants. 2020 Mar/Apr;35(2):423-431. doi: 10.11607/jomi.7869. PMID 32142580